CLINICAL TRIAL: NCT00766077
Title: Bone Geometry, Strength, and Biomechanical Changes in Runners With a History of Stress Fractures
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Laurie Moyer-Mileur Ph.D., R.D., University of Utah
Other Study IDs: 29496
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Stress Fractures; Bone Geometry; Bone Strength; Biomechanical Changes
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Stress fractures are a common and debilitating injury for a variety of athletes however current evidence does not clearly allow easy prediction of athletes at risk for a first fracture. Animal and some preliminary human evidence suggest that assessment of bone strength, muscle size and running mechanics may be primary risk factors for stress fractures. The investigators study will help determine which, if any, of these modifiable risk factors could help identify athletes at risk for stress fracture.

Competitive female distance runners will be recruited for this study. Participants will placed into a stress fracture or control group based on stress fracture history. Dual energy x-ray absorptiometry (DXA) and peripheral Quantitative Computed Tomography (pQCT) will be used to assess bone structure and strength. Running mechanics will be assessed during a 30-40 minute fatiguing run. A treadmill with an embedded force plate and high speed video will be used to assess changes in running mechanics throughout the run.

The purpose of this project will be to

1. explore differences in volumetric bone mineral density (vBMD), bone geometry, and muscle cross sectional area (MCSA) using pQCT
2. explore changes in load (GRFs) and running mechanics that occur during a fatiguing run in runners with and without a history of stress fracture.

DETAILED DESCRIPTION:
Stress fractures are among the most prevalent sports injuries, particularly in sports involving running, jumping, and repetitive cyclic loading. Stress fractures have been diagnosed in as many as 20% of athletes. The highest prevalence of stress fractures among athletes is reported in members of track and field teams with rates from 10-31% (22). Stress fractures are also a common occurrence in military basic training. U.S. military reports from the recruit populations indicate an incidence rate of 0.2 to 4% in men, and 1 to 7% in women (1).

Due to the prevalence of stress fractures in the military and athletic population, as well as the costly nature of the injury in terms of recovery time, it is important to understand the causative factors and the means by which these factors relate and interact (25, 29) . The most commonly studied and measured risk factors for stress fractures are surrogates of bone strength-particularly bone mineral density. Although several previous studies have explored the relationship of areal bone mineral density (aBMD, g/cm2) to stress fractures, the findings remain controversial (6, 7, 9, 12, 17, 28). A majority of these studies have used dual energy x-ray absorptiometry (DXA) and aBMD as the assessment of bone strength. DXA is limited in its 2-dimensional assessment of a 3-dimensional bone and is also unable to distinguish between different types of bone(13, 30). Given the limitations of DXA imaging, measuring bone properties using peripheral Quantitative Computed Tomography (pQCT) may shed light on inconsistencies found in the current literature. Peripheral QCT is a 3-dimensional imaging technique that allows for measurement of both trabecular and cortical volumetric bone density, bone geometry (total area, cortical area), and estimates of bone mechanical strength (i.e. cross-sectional moment of inertia and section modulus) which better represent a bones mechanical competence (26, 31).

With any fracture, a bone will fail only if the load on the bone is higher than the strength of that bone. In the case of stress fractures, it has been suggested that those at risk for stress fracture may alter biomechanics with fatigue such that strain on bone is increased with fatigue causing an increase in microdamage and ultimate fracture. Research measuring kinetic and kinematic variables has shown changes in GRFs (10, 11, 16, 19, 21), strain magnitude, strain rate, strain distributions (8, 14, 15, 24), and landing strategies after the onset of muscle fatigue in healthy individuals. It has also been shown that when muscles are fatigued, their ability to absorb impact forces during landing, their internal timing ability between functioning muscle groups, and ability to counter bending moments is decreased (2-5, 18, 20, 23). It has been hypothesized that runners who are ineffective at altering movement kinematics experience greater increases in loading rates and impact magnitudes, making them more susceptible to injury than runners who are able to make appropriate alterations (16). However, the majority of these studies have been conducted during resting conditions and in athletes with no history of injury. No previous studies to our knowledge have adequately characterized the change in biomechanics during a fatiguing run in athletes with and without a history of stress fracture.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be competitive female distance runners between the ages of 18-35.
* Athletes must currently be healthy, have been training for a minimum of 5 years and running 25 or more miles per week during their competitive season.

Exclusion Criteria:

* Participants will be excluded if they currently have a known chronic health problem, currently have a stress fracture or lower limb injury, currently have or have had an eating disorder, are on medication known to influence bone density and/or bone metabolism, or are pregnant. A pregnancy test will be administered to all female participants prior to any pQCT or DXA scans.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants must be competitive female distance runners between the ages of 18-35. Athletes must currently be healthy, have been training for a minimum of 5 years and running 25 or more miles per week during their competitive season.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Mileur, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States